CLINICAL TRIAL: NCT01781975
Title: Safety and Efficacy of Imatinib for Preserving Beta-Cell Function in New-Onset Type 1 Diabetes Mellitus
Brief Title: Imatinib Treatment in Recent Onset Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Stephen E. Gitelman, Director, Pediatric Diabetes Program, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-2013-6
Record Dates: First submitted 2013-01-17; First posted 2013-02-01 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type I; Diabetes Mellitus, Insulin-Dependent, 1; Type 1 Diabetes Mellitus; Insulin-Dependent Diabetes Mellitus 1; IDDM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib Mesylate (Experimental): 400 mg imatinib given once daily basis.
  Interventions: Drug: Imatinib Mesylate
- Placebo (Placebo Comparator): Placebo given once daily basis.
  Interventions: Drug: Placebo (For imatinib mesylate)

INTERVENTIONS:
Drug: Imatinib Mesylate
  Other Names: GLEEVEC; Glivec
  Arms: Imatinib Mesylate
Drug: Placebo (For imatinib mesylate)
  Arms: Placebo

SUMMARY:
Type 1 diabetes mellitus (T1DM) results from the autoimmune destruction of insulin-producing ß cells. Although exogenous insulin is widely available, it is not possible for affected individuals to consistently achieve euglycemia with current technology, and thus they are at risk for devastating long-term complications. This phase II study is designed to evaluate the safety and efficacy of imatinib mesylate as a novel therapy for new-onset T1DM. Imatinib is a first-in-class tyrosine kinase inhibitor.

This study will explore the potential role of short-term therapy with imatinib to induce tolerance and possibly lead to a durable long-term remission of T1DM.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive either imatinib mesylate or placebo daily.

All participants randomized into this study will be seen at a study site for a follow-up evaluation, 2 weeks and 4 weeks after randomization, and every month month thereafter for the first year. Participants will come in for a visit ever 6 months for the second year.

At the study visits, participants will undergo assessments of their insulin production, immunologic status, and overall health. Subjects will be followed until the conclusion of the study. The trial is expected to last approximately 2-4 years or until the required amount of information is gathered.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 12-45 years of age who meet the ADA standard T1DM criteria1. Positive for at least one islet cell autoantibody. Initial enrollment will be for subjects ages 18-45, with the goal to lower the age down to 12 upon acceptable safety review and prospect of benefit for this initial older cohort.
* Diagnosis of T1DM within 100 days of Visit 0.
* Peak stimulated C-peptide level >0.2 pmol/mL following an MMTT.
* Participants of childbearing age who are sexually active must agree to use an effective form of birth control (e.g., barrier method, oral contraception, or surgery). For females, these contraceptive measures must be maintained throughout the study; for males these measures must be followed for a minimum of 3 months after discontinuation of imatinib therapy.

Exclusion Criteria:

* Prior history of any significant cardiac disease such as congestive heart failure, myocardial infarction, arrhythmia, or structural defects or suspicion thereof.
* Leukopenia (<3,000 leukocytes/μL), neutropenia (<1,500 neutrophils/μL), or thrombocytopenia (<125,000 platelets/μL).
* Low Hemoglobin (baseline hemoglobin below lower limit of normal)
* Prior history of anaphylaxis, angioedema or serious cutaneous drug reactions
* Any sign of significant chronic active infection (e.g., hepatitis, tuberculosis, EBV, CMV, or toxoplasmosis), or screening laboratory evidence consistent with a significant chronic active infection (such as positive for HIV, PPD, or HBSAg). Significant acute infections must be resolved before treatment may commence, e.g., acute respiratory tract, urinary tract, or gastrointestinal tract infections.
* Anticipated ongoing use of diabetes medications other than insulin that affect glucose homeostasis, such as metformin, sulfonylureas, thiazolidinediones, glucagon-like peptide 1 (GLP-1) mimetics, dipeptidyl peptidase IV (DPP-IV) inhibitors, or amylin.
* Prior or current treatment that is known to cause a significant, ongoing change in the course of T1DM or immunologic status, including high-dose inhaled, extensive topical or systemic glucocorticoids.
* Evidence of liver dysfunction, with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 times the upper limit of normal persistent for 1 week or greater.
* Evidence of renal insufficiency as indicated by serum creatinine > 1.2 times the upper limit of normal and confirmed in a repeat test at least one week apart. Evidence of clinically significant metabolic bone disease (except adequately treated rickets).
* Females who are pregnant at the time of screening or unwilling to defer pregnancy during the 24-month study period.
* Prior treatment with imatinib or related tyrosine kinase inhibitor.
* Unable to avoid medications that affect CYP3A4: either inducers that may decrease imatinib levels, or inhibitors that may increase drug concentrations. (Refer to section 1.5.1.12 for a complete list of inducers and inhibitors.)
* Height standard deviation score ≥2 standard deviations below mean
* Any sign of QT prolongation on Visit -1 noted on ECG (> 450 ms in males and > 470 ms in females)
* Known coagulation disorders or use of anticoagulants
* Current and anticipated on-going treatment with drugs that may increase or decrease imatinib plasma concentrations (CYP3A4 family inhibitors or inducers) or drugs that may have their plasma concentration altered by imatinib (drugs metabolized by CYP3A4/5 and CYP2D6).
* Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Gitelman, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (8):
  - University of California-San Francisco, San Francisco, California
  - Barbara Davis Center, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
- Walter and Eliza Hall Institute of Medical Research, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Gitelman SE, Bundy BN, Ferrannini E, Lim N, Blanchfield JL, DiMeglio LA, Felner EI, Gaglia JL, Gottlieb PA, Long SA, Mari A, Mirmira RG, Raskin P, Sanda S, Tsalikian E, Wentworth JM, Willi SM, Krischer JP, Bluestone JA; Gleevec Trial Study Group. Imatinib therapy for patients with recent-onset type 1 diabetes: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2021 Aug;9(8):502-514. doi: 10.1016/S2213-8587(21)00139-X. Epub 2021 Jun 29. PMID 34214479
- [Derived] Robertson MA, Padgett LR, Fine JA, Chopra G, Mastracci TL. Targeting polyamine biosynthesis to stimulate beta cell regeneration in zebrafish. Islets. 2020 Sep 2;12(5):99-107. doi: 10.1080/19382014.2020.1791530. Epub 2020 Jul 25. PMID 32715853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2013 to May 2016 at 9 clinical sites (8 US, 1 Australia)
Groups:
- Imatinib Mesylate: 400 mg imatinib given once daily basis.
  Imatinib Mesylate
- Placebo: Placebo given once daily basis.
  Placebo (For imatinib mesylate)
Period: Overall Study
Arm/Group | Imatinib Mesylate | Placebo
Started | 45 | 22
Treatment Period | 44 | 22
Follow-Up Period | 43 | 21
Completed | 43 | 21
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate | Placebo | Total
Number analyzed (Participants) | 45 | 22 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 22 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (7.2) | 26.2 (6.6) | 27 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 27 | 10 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 43 | 19 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 21 | 65
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 18 | 54
  Australia | 9 | 4 | 13
Number of Autoantibodies Positive [Count of Participants; unit: Participants]
  1 | 8 | 4 | 12
  2 | 8 | 4 | 12
  3 | 12 | 1 | 13
  4 | 8 | 6 | 14
  5 | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Stimulated C-peptide Curve (AUC) Mean Over the First 2 Hours of a 4 Hour Mixed Meal Tolerance Test at the 1 Year Visit
Description: The primary outcome of each participant is the area under the stimulated c-peptide curve (AUC) mean based on data collected at time 0 to 2 hours of a 4-hour mixed meal tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30, 60, 90, and 120 minutes. The term "AUC mean" comes from the mean value theorem in calculus. It is the value on the scale of the y-axis that is equal to the AUC divided by the range on the x-axis (in this case 120 minutes).
Time Frame: Visit 9 (Week 52) at 0, 15, 30, 60, 90, 120 minutes post-dose
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
nmol/L | 0.834 (0.446) | 0.775 (0.278)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.048, ANCOVA; ANCOVA = 0.0616, 90% CI 2-sided [0.00176 to 0.121], Standard Error of Mean 0.0364

2. Secondary Outcome: Area Under the Stimulated C-peptide Curve (AUC) Mean Over 4 Hours at 24 Months
Description: Area under the MMTT-stimulated peak, 4 hour C-peptide AUC mean at week 104. The units are reported as nano-moles/Liter because this is AUC mean (the AUC is divided by the time internal so that the units return to the c-peptide units of measure).
Time Frame: Visit 13 (Week 104)
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
nmol/L | 0.472 [0.355 to 0.599] | 0.389 [0.255 to 0.538]

3. Secondary Outcome: Change in HbA1c Levels Over Time
Description: Change in HbA1c levels from Week 52 to Week 104
Time Frame: Visit 9 (Week 52) and Visit 13 (Week 104)
Measure: Mean (95% Confidence Interval); unit: percentage of HbA1c level
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
percentage of HbA1c level
  Week 52 | 6.33 [6.02 to 6.66] | 6.51 [6.03 to 7.02]
  Week 104 | 6.44 [6.09 to 6.81] | 7.03 [6.42 to 7.69]

4. Secondary Outcome: Change in Insulin Dose (Units/kg) Over Time
Description: Assess insulin use in units per kilogram body weight per day at weeks 52 and 104.
Time Frame: Visit 9 (Week 52) and Visit 13 (Week 104)
Measure: Mean (95% Confidence Interval); unit: Units per Kg
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
Units per Kg
  Week 52 | 0.307 [0.24 to 0.379] | 0.413 [0.279 to 0.56]
  Week 104 | 0.389 [0.315 to 0.467] | 0.488 [0.353 to 0.637]

5. Secondary Outcome: Number of Severe Hypoglycemic Events
Description: Major hypoglycemic events occurring from randomization at weeks 0, 52 and 104.
Time Frame: Visit 0 (Week 0), Visit 9 (Week 52), and Visit 13 (Week 104)
Measure: Number; unit: events
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
events | 2 | 3

6. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events that were reported throughout the study.
Time Frame: Adverse Events will be assessed at Visit 0 (week 0), Visit 1 (Week 2), Visit 2 (Week 4), and every month thereafter.
Measure: Number; unit: events
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 45 | 22
events | 172 | 28

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events that were not considered Serious Adverse Events (SAE) were monitored/assessed without regard to the specific Adverse Event Term so the categories they belong to are provided below.
Arm/Group | Imatinib Mesylate | Placebo
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/22
Serious Adverse Events (participants affected / at risk) | 8/45 | 3/22
Other Adverse Events (participants affected / at risk) | 23/45 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=45) | Placebo (N=22)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Fluid in Lungs (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Diabetes ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (3) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Respiratory Acidosis, Likely secondary to hypo ventilation in setting of severe lethargy
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prutitus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Axillary Abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=45) | Placebo (N=22)
Infections and infestations (Infections and infestations) | 12 (26) | 4 (9)
Eye disorders (Eye disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Nervous system disorders (Nervous system disorders) | 4 (4) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (13) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 (11) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 5 (9) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 4 (6) | 0 (0)
General disorders & administration site condt'ns (General disorders) | 2 (2) | 0 (0)
Investigations (Investigations) | 10 (18) | 2 (4)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 3 (5) | 2 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 (7) | 0 (0)
Endocrine disorders (Endocrine disorders) | 4 (45) | 1 (2)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
FDA did not approve for hold on enrollment of pediatric population to be lifted; only adult population was recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT01781975/Prot_SAP_000.pdf